CLINICAL TRIAL: NCT02944929
Title: Randomised Controlled Trial to Evaluate the Effect of a Self-rehabilitation Program in Addition to Usual Treatment for Spasticity (Repeated Botulinum Toxin Injections and Physiotherapy) on Impairment and Activity Limitation in Patients With Spastic Hemiparesis Following Stroke
Brief Title: The Effect of a Self-rehabilitation Program in Addition to Usual Treatment for Spasticity on Impairment and Activity Limitation in Patients With Spastic Hemiparesis Following Stroke
Acronym: ADJU-TOX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P150907
Record Dates: First submitted 2016-09-14; First posted 2016-10-26 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Spastic Hemiparesis
Keywords: Spastic hemiparesis; Stroke; Self-rehabilitation; Botulinum Toxin Injections
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-rehabilitation program (Experimental): Self-rehabilitation program + standard medical care (BTI + conventional physiotherapy)
  Interventions: Other: Self-rehabilitation program
- Control arm (No Intervention): Arm with standard medical care ( BTI + conventional physiotherapy) without self-rehabilitation program

INTERVENTIONS:
Other: Self-rehabilitation program — The self-rehabilitation program will be based on muscle stretching, strengthening and task oriented exercises. For each patient, two exercises will be selected by the therapist for each of these 3 domains (total of 6 exercises) from a list of 50 exercises.
  Arms: Self-rehabilitation program

SUMMARY:
The addition of a self-rehabilitation program to repeated Botulinum Toxin Injections (BTI) and usual physiotherapy should increase the proportion of patients who attain their Primary Treatment Goal (impairments and function) more than usual care (involving repeated Botulinum Toxin Injections and conventional physiotherapy), in post stroke out-patients with spasticity.

DETAILED DESCRIPTION:
Stroke affects 150 000 persons in France each year. Most patients have activity limitations because of the resulting motor deficit and spasticity. Autonomy in activities of daily living is reduced.

The principal treatment for focal spasticity is currently intramuscular botulinum toxin injection (BTI).

BTI is classically combined with only 2 to 3 sessions of out-patient physiotherapy per week. This is mainly because of a lack of out-patient therapists. However, this amount of therapy is insufficient and does not follow current literature which shows that the intensity of physiotherapy affects the recovery of impairment and activity. This gap in our health system could be filled by a self-rehabilitation program in addition to physiotherapy.

Recent studies have shown that self-rehabilitation following BTI could significantly improve activity limitation (Roche et al, 2014 ; Sun et al 2010).

The addition of a self-rehabilitation program to BTI and usual out-patient physiotherapy could thus increase the effects of BTI on impairment and activity limitation in patients with spastic hemiparesis following stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged between 18 to 75 years.
2. Adult patient under guardianship with consent obtained and the legal guardian's authorisation obtained.
3. Single stroke having occurred more than 6 months before (previous TIA is accepted).
4. Capable of understanding instructions and participating in the definition of a therapeutic goal (Boston Diagnostic Aphasia Examination (BDAE) < 3).
5. Having previously undergone BTI. The last injection must have been performed at least 4 months prior to inclusion.
6. Affiliation to the French social security regime or a similar regime.
7. Patient (or the legal guardian if under guardian adult patient) has signed the informed consent form.

Exclusion Criteria:

1. Patients who are unwilling to participate in the study. For the one under guardianship, the refusal of the patient will be the final decision even if the guardian is willing to participate.
2. Subjects who are unlikely to adhere to the study an/or poor adherence anticipated by the investigator.
3. Un-controlled progressive pathology.
4. Osteoarticular lesion which contraindicates part of the rehabilitation involved in the study.
5. Patients with other interventions planned prior to the end of the study period (orthosis, surgery etc.).
6. Surgery to the treated limb less than 6 months previously.
7. Pregnant woman.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-01-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of Goal Attainment Scaling (GAS). | 6 months
  The percentage of patients who attain their Primary Treatment Goal determined using Goal Attainment Scaling (GAS) at each visits and in both groups.

SECONDARY OUTCOMES:
Assessment of the Functional Independence Measure (FIM) | 6 months
Assessment of Hemispatial neglect | 6 months
Quality of life questionnaire | 6 months
Assessment of slight deficits according MOCA scale (Montréal Cognitive Assessment) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Roche, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Raymond Poincaré, Garches, France

REFERENCES:
- [Derived] Bonnyaud C, Gallien P, Decavel P, Marque P, Aymard C, Pellas F, Isner ME, Boyer FC, Muller F, Daviet JC, Dehail P, Perrouin-Verbe B, Bayle N, Coudeyre E, Perennou D, Laffont I, Ropers J, Domingo-Saidji NY, Bensmail D, Roche N; ADJU-TOX Study Group. Effects of a 6-month self-rehabilitation programme in addition to botulinum toxin injections and conventional physiotherapy on limitations of patients with spastic hemiparesis following stroke (ADJU-TOX): protocol study for a randomised controlled, investigator blinded study. BMJ Open. 2018 Aug 30;8(8):e020915. doi: 10.1136/bmjopen-2017-020915. PMID 30166290